CLINICAL TRIAL: NCT00297076
Title: A Phase III, Randomized, Double-Blind, Placebo-Controlled, Multicenter, Parallel Group Study to Compare the Efficacy and Safety of GW873140 400mg BID in Combination With a Ritonavir-Containing Optimized Background Therapy (OBT) Regimen Versus Placebo Plus OBT Over 48 Weeks.
Brief Title: Chemokine Coreceptor 5 (CCR5) Antagonist GW873140 In R5-Tropic Treatment-Experienced HIV-Infected Subjects
Status: Terminated | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Study Director, GSK
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CCR104456
Record Dates: First submitted 2006-02-24; First posted 2006-02-27 (Estimated); Last update posted 2009-05-18 (Estimated); Status verified 2009-05

CONDITIONS: HIV Infection
Keywords: HIV-1; GW873140; CCR5 antagonist; experienced; Treatment Experienced
MeSH Terms: conditions — HIV Infections | interventions — aplaviroc

INTERVENTIONS:
Drug: GW873140

SUMMARY:
The purpose of this study is to evaluate the safety and efficacy of the CCR5 antagonist GW873140 or placebo in combination with an optimized background regimen in treatment-experienced HIV-infected subjects with R5-tropic virus

ELIGIBILITY:
Inclusion Criteria:

* The following are study specific eligibility criteria. In addition to these criteria, investigators must exercise clinical discretion regarding selection of appropriate study subjects, taking into consideration any local treatment practices or guidelines.

A subject will be eligible for inclusion in the CCR104456 protocol only if all of the following criteria apply:

* HIV-1 infected subjects aged 18 years or older. All subjects participating in this study should be counseled on the practice of safe sex throughout the study. Females must fall into one of the following categories:

Non-childbearing potential: defined as women who are surgically sterile or post-menopausal, the latter indicated by history of no menses for a minimum of one year prior to the date of the screening visit; Childbearing potential: has a negative pregnancy test result (-human chorionic gonadotropin; -HCG) within 35 days prior to administration of investigational product (Day 1) and agrees to use a proven double barrier method of contraception (e.g. spermicide + condom) during the study period (through follow-up). Hormonal contraceptives will not be considered sufficient forms of contraception for this study.

* Screening plasma HIV-1 RNA ≥5000copies/mL (from CCR104627 protocol). There are no CD4 cell count entry restrictions, however investigators must exercise clinical discretion regarding selection of appropriate study subjects, taking into consideration any local treatment practices or guidelines regarding CD4 cell count and HIV-1 RNA.
* Total prior antiretroviral experience of at least three months and documented genotypic or phenotypic resistance to at least one compound in each of the following classes of antiretrovirals: NRTIs (includes NtRTI TDF), NNRTIs, and PIs. Resistance mutations must be at least one major mutation according to the current International AIDS Society-USA Drug Resistance Mutations Group (refer to study reference manual [SRM]). Resistance testing may be current (e.g. screening results) and/or historical with verifiable documentation in source documents.
* R5-tropic virus according to viral tropism assessment at screening in CCR104627 protocol.
* Current receipt of an unchanged "pre-study" ART regimen (i.e., unchanged medications and doses) for at least four weeks prior to screening in CCR104627 protocol; this pre-study regimen may be no ART. Subjects must remain on this regimen until randomization (Day 1).
* Subjects must be able to receive a RTV-boosted PI as part of their OBT regimen. Due to the possibility of randomization to the placebo arm, investigators should consider subjects for enrollment whose treatment history and resistance testing results suggest that an OBT regimen can be constructed which would be anticipated to provide the best possible virological response and clinical benefit for each subject. The drugs in the OBT regimen will be chosen from the locally available antiretrovirals and must consist of between three and six drugs, one of which must be a RTV-boosted PI. Use of investigational PIs which become available through expanded-access or similar programs during the conduct of this study must be authorized by the Sponsor prior to use in OBT regimen.
* Ability to understand and comply with protocol requirements, instructions and protocol-stated restrictions.
* Signed and dated written informed consent prior to initiation of pre-baseline study procedures.

Exclusion Criteria:

A subject will not be eligible for inclusion in the CCR104456 protocol if any of the following criteria apply:

* Plasma sample tests as R5/X4 (dual or mixed)-tropic, X4-tropic only, or non-phenotypeable based on viral tropism assessment at screening in protocol CCR104627.
* Any acute laboratory abnormality at screening which, in the opinion of the investigator, should preclude the subject's participation in the study of an investigational compound. Any Grade 4 laboratory abnormality at screening will exclude a subject from study participation unless the investigator can provide a compelling explanation for the laboratory result(s) and has the assent of the Sponsor.
* Subjects that make any changes to their ART regimen during the period beginning four weeks prior to screening (protocol CCR104627) until Day 1.
* Significant blood loss (≥500mL) within 56 days prior to screening in CCR104627 protocol.
* Pregnant women or women who are breastfeeding.
* Previous participation in an experimental drug and/or vaccine trial(s) within 30 days or 5 half-lives, or twice the duration of the biological effect of the experimental drug or vaccine - whichever is longer, prior to screening for the study.
* Subjects with any prior receipt of an investigational CCR5 or CXCR4 antagonist are excluded.
* Any clinically significant finding on screening or baseline ECG. Specifically, subjects with any repolarization delay (resting QTcB interval >450msec at the screening or baseline [mean of triplicate values] visit) will be excluded. Subjects with a history of additional risk factors for torsade de pointes (e.g., heart failure, chronic and/or recurrent hypokalemia) will also be excluded.
* History of clinically relevant pancreatitis or hepatitis within the previous 6 months. Asymptomatic individuals with chronic hepatitis B (HBV) or hepatitis C virus (HCV) infection will not be excluded, however investigators should carefully assess if antiviral therapy specifically for HBV or HCV infection is required; subjects who are anticipated to require such therapy during the study should be excluded.
* Any condition which, in the opinion of the investigator, may interfere with the subject's ability to comply with the dosing schedule and/or protocol evaluations (including alcohol or drug abuse) or which might compromise the safety of the subject.
* Any evidence of active CDC Class C conditions or opportunistic infections. Subjects on stable, anti-infective treatment or prophylaxis regimen are allowed in the study provided the therapy is not specifically prohibited.
* Any condition which, in the opinion of the investigator, might interfere with the absorption, distribution, metabolism, or excretion of the drug.
* History of a drug or other allergy which, in the opinion of the investigator, contraindicates the subject's participation in the study or known hypersensitivity to any study medication or excipients.
* Treatment with radiation therapy or cytotoxic chemotherapeutic agents within 30 days of investigational product administration or anticipated need for such treatment during the study.
* Current severe illness, including liver and renal failure, major organ allograft, malignancy requiring parenteral chemotherapy that can not be discontinued for the duration of the trial, or any other conditions which would make the subject unsuitable for the study. Subjects with basal cell carcinoma of the skin, in situ carcinoma of the cervix, or non-disseminated stable Kaposi's sarcoma may be included in the trial.
* Use of systemic immunosuppressants and/or immunomodulators within 30 days prior to study Day 1. Systemic corticosteroids at replacement doses (e.g. 10mg/day prednisone or equivalent) are permitted.
* Anticipated continued need for prescription or over-the-counter (OTC) medications that are on the prohibited medication list within 30 days prior to study Day 1.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 406
Dates: Start 2005-07; Primary Completion 2007-10 (Estimated); Study Completion 2007-10 (Estimated)

PRIMARY OUTCOMES:
HIV viral load response at 24 and 48 weeks as measured by proportion of subjects with undetectable viral load, change from baseline over time, proportion of subjects with 1.0 log drop, and time to virologic failure.

SECONDARY OUTCOMES:
Safety and tolerability, change in T-cell count, disease progression, viral resistance,tropism at failure, pharmacokinetics, health outcomes, and adherence will be determined over 24 and 48 weeks. Liver tests will be done every 2 weeks for 24 weeks.
Proportion of subjects with plasma HIV-1 RNA <400copies/mL at Week 24 and 48 based on the outcomes from the TLOVR algorithm.

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Ph.D., Study Director — GlaxoSmithKline
Locations (4):
- Germany (4):
  - GSK Investigational Site, Frankfurt am Main, Hesse
  - GSK Investigational Site, Hanover, Lower Saxony
  - GSK Investigational Site, Düsseldorf, North Rhine-Westphalia
  - GSK Investigational Site, Berlin, State of Berlin